CLINICAL TRIAL: NCT02108340
Title: Comparative Study of Microwave Radiometry and Ultrasonography for the Diagnosis of Acute Appendicitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Toutouzas, Assistant Professor of Surgery, Hippocration General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ΕΣ 45/19-9-2013
Record Dates: First submitted 2014-04-02; First posted 2014-04-09 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Appendicitis
Keywords: Appendicitis; Diagnosis; Microwave radiometry; Ultrasonography
MeSH Terms: conditions — Appendicitis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Microwave radiometry (Experimental): Patients diagnosed with acute appendicitis will undergo a measurement of the temperature of the appendix with the use of microwave radiometry in a room temperature of 20 -24 degrees celsius.
  Interventions: Procedure: Microwave radiometry

INTERVENTIONS:
Procedure: Microwave radiometry — Microwave radiometry of the right lower quadrant in a room temperature of 20-24 degrees celsius, in order to record changes in the temperature of the inflamed appendix.

SUMMARY:
This study will evaluate the use of microwave radiometry in a population of patients diagnosed with acute appendicitis and treated with appendectomy. The main purpose of the study is to report the results of microwave radiometry as a diagnostic tool in acute appendicitis and compare those results with the commonly used ultrasonography.

DETAILED DESCRIPTION:
Patients diagnosed with acute appendicitis from the emergency department of Hippocration General Hospital and treated with appendectomy will be evaluated with microwave radiometry for changes in the temperature of the appendix before its removal.

Subsequently, the results of microwave radiometry for the patients confirmed by the histopathology report to have acute inflammation of the appendix, will be compared with those of the ultrasonography used for the diagnosis of acute appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of appendicitis
* Surgical removal of appendix
* Pathological confirmation of appendicitis

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Appendix Temperature | Baseline
  Microwave radiometry will assess the temperature of the appendix for the patients diagnosed with appendicitis before they undergo surgical removal of the appendix.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos G. Toutouzas, MD, PhD, Study Chair — Hippocration General Hospital; Evagelia Stamouli, MD, Principal Investigator — Hippocration General Hospital
Locations (1):
- Hippocration General hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Toutouzas K, Grassos C, Drakopoulou M, Synetos A, Tsiamis E, Aggeli C, Stathogiannis K, Klettas D, Kavantzas N, Agrogiannis G, Patsouris E, Klonaris C, Liasis N, Tousoulis D, Siores E, Stefanadis C. First in vivo application of microwave radiometry in human carotids: a new noninvasive method for detection of local inflammatory activation. J Am Coll Cardiol. 2012 May 1;59(18):1645-53. doi: 10.1016/j.jacc.2012.01.033. PMID 22538335
- [Background] Arunachalam K, Maccarini PF, De Luca V, Bardati F, Snow BW, Stauffer PR. Modeling the detectability of vesicoureteral reflux using microwave radiometry. Phys Med Biol. 2010 Sep 21;55(18):5417-35. doi: 10.1088/0031-9155/55/18/010. Epub 2010 Aug 25. PMID 20736499
- [Background] Toutouzas K, Grassos H, Synetos A, Drakopoulou M, Tsiamis E, Moldovan C, Agrogiannis G, Patsouris E, Siores E, Stefanadis C. A new non-invasive method for detection of local inflammation in atherosclerotic plaques: experimental application of microwave radiometry. Atherosclerosis. 2011 Mar;215(1):82-9. doi: 10.1016/j.atherosclerosis.2010.12.019. Epub 2010 Dec 23. No abstract available. PMID 21256490
- [Background] Hassan AM, El-Shenawee M. Review of electromagnetic techniques for breast cancer detection. IEEE Rev Biomed Eng. 2011;4:103-18. doi: 10.1109/RBME.2011.2169780. PMID 22273794